CLINICAL TRIAL: NCT06668233
Title: Neurocognitive Disorders in Children with Congenital Heart Disease
Brief Title: Neurologocal Symptoms in CHD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Salah Mahmoud Ahmed, doctor, Assiut University
Other Study IDs: neurologocal symptoms in CHD
Record Dates: First submitted 2024-09-22; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-09

CONDITIONS: Neurological Disorders
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children from 3 years to 18 years with congenital heart disease
  Interventions: Radiation: CT; Radiation: CT scan

INTERVENTIONS:
Radiation: CT — CT Brain
Radiation: CT scan — Neuroimaging in case with delayed development , focal neurological symptoms or seziures

SUMMARY:
The aim of the study is to determine neurological and cognitive disorders in children with congenital heart disease for early diagnosis and treatment

DETAILED DESCRIPTION:
Congenital heart defects are significant structural abnormalities affecting the heart and major intrathoracic vessels. They are among the most common birth defects, constituting about one-third of all major congenital anomalies. Many of these defects necessitate surgical intervention during early childhood. Advances in surgical techniques have significantly improved survival rates for patients with congenital heart disease (CHD). However, a variety of systemic complications have become more apparent, including issues affecting the cardiac, pulmonary, gastrointestinal, neurological, and nephrological systems (Walaa El Naga et al., 2022).

Neurological complications greatly contribute to morbidity and mortality in pediatric CHD patients, significantly impacting their neurodevelopmental outcomes. Various studies indicate that up to 30% of children with congenital heart disease (CHD) experience neurological complications. Seizures are the most frequently reported neurological complication, accounting for approximately 70% of cases with neurological sequelae (Aly El Kazaz et al., 2022).

Also Neuropsychological studies of children with complex CHD reveal distinct deficits in intelligence, cognitive performance, executive function, language skills, visuospatial abilities, and attention. (Guo et al., 2021). Recognizing the long-term consequences of accumulated brain injury underscores the importance of identifying and minimizing early insults. (Le H.Sterling et al., 2021) The recognized neurodevelopmental challenges faced by children with CHD prompted the American Heart Association to recommend routine neurodevelopmental evaluations for high-risk patients with CHD. According to the American Heart Association, the initial visit, conducted before 12 months of age, should include a neuromotor examination assessing muscle tone, primitive and deep tendon reflexes, sensory status, and gross motor skills. Although many children with CHD now undergo these recommended neurological examinations, the examinations and their outcomes have not been thoroughly described. Additionally, factors predicting abnormal neurological examination results have not been identified. Enhancing our understanding of the findings from these routinely recommended evaluations will improve the detection of abnormalities, thereby optimizing support for children with CHD and their families.(Le Samantha butler et al., 2023).

ELIGIBILITY:
Inclusion Criteria:

- Children from 3 years to 18 years with congenital heart disease

Exclusion Criteria:

* New born infants. Children with normal heart. Children with chromosomal or metabolic disease.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 3 years to 18 years with congenital heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The aim of the study is to determine neurological and cognitive disorders in children with congenital heart disease for early diagnosis and treatment. | one year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butler SC, Sadhwani A, Rofeberg V, Cassidy AR, Singer J, Calderon J, Wypij D, Newburger JW, Rollins CK; Cardiac Neurodevelopmental Program at Boston Children's Hospital Group. Neurological features in infants with congenital heart disease. Dev Med Child Neurol. 2022 Jun;64(6):762-770. doi: 10.1111/dmcn.15128. Epub 2021 Dec 18. PMID 34921736